CLINICAL TRIAL: NCT04448574
Title: Chest Wall Deformities in Children - Epidemiological Data
Status: Completed | Type: Observational
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Principal Investigator, Dr. med. Julian Trah, Medical Doctor, Universitätsklinikum Hamburg-Eppendorf
Other Study IDs: CWD2019
Record Dates: First submitted 2020-06-24; First posted 2020-06-26 (Actual); Last update posted 2021-12-07 (Actual); Status verified 2021-12

CONDITIONS: Chest Wall Deformity; Funnel Chest
MeSH Terms: conditions — Funnel Chest

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Chest Wall Deformities Questionaire — Questionaire about epidemiological data was sent to Patients and families

SUMMARY:
Pectus excavatum (PE) or funnel breast is the most common congenital deformity of the chest wall, which occurs in about 1 in 400 births with a boy to girl ratio of 4: 1 to 3: 1. The etiology of PE is largely undefined, but there are numerous indications that genetic factors play a role in the development of PE. Up to 40% of patients report affected family members with similar congenital deformities. In many families, PE follows a pattern that would be compatible with an autosomal dominant or recessive pattern of inheritance. The data on the frequent occurrence of PE in family members fluctuate greatly and only a few genes associated with a PE have been identified so far.

DETAILED DESCRIPTION:
Previous studies suggest that sulfation of proteoglycans plays a crucial role in the normal development of cartilage and bone and could therefore be crucial in the genesis of the disease. The main catalytic machinery responsible for the biosynthesis and breakage of sulfate esters in the proteoglycans consists of various enzymes and transporters. Mutations in Sphingosine Kinase 1 (SK1) and Sphingosine Kinase 2 (SK2) genes that encode the transmembrane transporters of sulfate or enzymes that are involved in 3'-phosphoadenosine 5'-phosphosulfate (PAPS) synthesis have been identified as the cause of several inherited diseases that all have skeletal system deformities.

Connections between chest wall deformities with syndromes (e.g. Marfan, Noonan), anomalies (e.g. Poland, Moebius) or associations (e.g. Cantrell Pentalogy, PHACE) are well known. In contrast, there have so far been hardly any genetic studies of the isolated congenital chest wall deformities. Epidemiological data are insufficient and only a few groups deal with the inheritance and the incidence of this disease when it occurs in isolation.

ELIGIBILITY:
Inclusion Criteria:

* . All patients who are in the Altona Children's Hospital or in the University Hospital Hamburg. Funnel breast, keel breast, sternal cleft
* . A signed declaration of consent from the parents or legal guardians is available
* . The patient has given a declaration of consent

Exclusion Criteria:

* Confirmation of another diagnosis associated with chest wall deformities:

  1. Marfan syndrome
  2. Noonan syndrome
  3. Poland syndrome
  4. Moebius syndrome
  5. Cantrell Pentalogy
  6. PHACE association

Ages: 6 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All patients who presented themselves in the study hospitals with the diagnosis of a chest wall deformity (funnel breast, keel breast, sternum cleft)
Sampling Method: Non-Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
familial accumulation of breast wall deformities Questionnaire | Through study completion, an average of 1 year

SECONDARY OUTCOMES:
Recording of clinical side effects on the familial accumulation of chest wall deformities | Through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - University Hospital Hamburg Eppendorf - Department of pediatric surgery, Hamburg
  - The Altona Children's Hospital, Hamburg

IPD SHARING:
Plan to Share IPD: No